CLINICAL TRIAL: NCT07128953
Title: The First Affiliated Hospital of Anhui University of Chinese Medicine
Brief Title: Study on the Mechanism of Zuoqing San Promoting Postoperative Wound Healing of Anal Fistula by Inhibiting ROS-dependent NETosis
Acronym: ZQS
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Heng Deng, The First Affiliated Hospital of Anhui University of Chinese Medicine, The Second Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024AH-97-01; 2023AH050848 (Other Grant/Funding Number: cientific Research Project of Colleges and Universities of Anhui Province)
Record Dates: First submitted 2025-07-17; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Anal Fistula
Keywords: Anal fistula
MeSH Terms: conditions — Rectal Fistula | interventions — Fumigation

STUDY DESIGN:
Intervention Model Description: Inclusion criteria**
  1. **Western medical diagnostic criteria** (refer to "Surgery for Anorectal Diseases" 2018 edition):
  * History of recurrent swelling and pus discharge around the anus;
  * Confirmed presence of fistula through preoperative MRI or ultrasound;
  * Undergone incisional surgery for anal fistula, with postoperative wound diameter ranging from 2 to 4 cm.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): ZQS
  Interventions: Drug: Solution of Zuoqing San for fumigation and washing of the postoperative wound of anal fistula
- control Group (Placebo Comparator): Control
  Interventions: Other: Equal-volume placebo inhalation rinse

INTERVENTIONS:
Drug: Solution of Zuoqing San for fumigation and washing of the postoperative wound of anal fistula — Left Qing San Decoction (25g of Cai Yin + 30g of Eucommia + 25g of Sophora flavescens + 25g of Anemarrhena asphodeloides + 15g of Lithospermum erythrorhizon, prepared in the Pharmacy Department of Anhui University of Traditional Chinese Medicine), add 1000mL of water, boil, then steam and wash the wound surface. The temperature is 40 ± 2℃. Do it once a day, for 15 minutes each time, for 7 consecutive days.
  Arms: Study Group
Other: Equal-volume placebo inhalation rinse — Equal-volume placebo inhalation rinse
  Arms: control Group

SUMMARY:
This study adopted a randomized, double-blind, placebo-controlled clinical trial design to evaluate the efficacy and safety of Zuoqing San fumigation and washing on the wound healing after anal fistula surgery.

DETAILED DESCRIPTION:
A total of 60 patients who underwent anal fistula surgery at the Second Affiliated Hospital of Anhui University of Chinese Medicine from September 2024 to March 2025 were included. They were randomly divided into the experimental group (treated with Left Qing San fumigation and washing) and the control group (treated with placebo fumigation and washing) at a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent swelling and pain, along with pus discharge around the anus;
* Preoperative MRI or ultrasound confirmed the presence of the fistula;
* Underwent incision of the anal fistula, with the postoperative wound diameter ranging from 2 to 4 cm.

Exclusion Criteria:

1. Inflammatory bowel disease (such as Crohn's disease) related anal fistula;
2. Complicated with severe dysfunction of heart, liver and kidney (ALT/AST > 2 times upper limit, Cr > 1.5 mg/dL);
3. Pregnant or lactating women;
4. Those who are known to be allergic to the components of Zuoqing San;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-08-02 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Wound healing time | From postoperative day 1 until wound healing is achieved (assessed daily during hospitalization and weekly after discharge, up to 8 weeks)
  The number of days from the day after the operation until the wound surface is completely covered by epithelium (as observed by the naked eye, there is no exudation, and upon palpation, the scar is smooth).

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui university of Chinese Medicine, Hefei, Anhui, China